CLINICAL TRIAL: NCT06349408
Title: A Phase 1 Study of IBI3001 in Participants With Unresectable, Locally Advanced or Metastatic Solid Tumors
Brief Title: IBI3001 in Participants With Unresectable, Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3001A101
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label: IBI3001 monotherapy (Experimental)
  Interventions: Drug: IBI3001

INTERVENTIONS:
Drug: IBI3001 — The provisional dose levels are planned to be evaluated, but it is possible for additional and/or intermediate dose levels to be added during the study.
  IBI3001 is proposed to be administered by intravenous infusion (IV)

SUMMARY:
This is a Phase 1 multicenter, multi-regional, open-label, first-in-human study of IBI3001 in participants with unresectable, locally advanced or metastatic solid tumors. The purpose of this study is to identify the MTD/RP2D of IBI3001, and to explore the preliminary efficacy of IBI3001.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants ≥ 18 years old;
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
3. Has an anticipated life expectancy of ≥ 12 weeks;
4. Adequate bone marrow and organ function:
5. At least 1 evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. for dose escalation , and 1 measurable lesion for dose expansion.
6. Has a documented (histologically- or cytologically-proven), unresectable, locally advanced or metastatic solid tumor that is refractory to or intolerable with standard treatment, or for which no standard treatment is available; participants who refuse standard therapy, or are able to suspend standard therapy without major risks.

Key Exclusion Criteria:

1. Progressed or refractory to an ADC that consists of an Exatecan derivative that is a topoisomerase I inhibitor or intolerable with an ADC that consists of Exatecan;
2. Plan to receive other antitumor therapy during the study excluding palliative radiotherapy for the purpose of symptom (like pain) relief that must also not have an impact on tumor assessment throughout the study;
3. Pyloric obstruction and/or persistent recurrent vomiting (≥ 3 times in 24 hours);
4. Gastrointestinal perforation and/or fistula within 6 months prior to first administration of the study drug, and not recovered after surgical treatment;
5. Known symptomatic central nervous system (CNS) metastases.
6. History of pneumonia requiring corticosteroids therapy, or history of clinically significant lung diseases; Uncontrolled diseases;
7. History of endotracheal or gastrointestinal stent implantation;
8. Ascites, pleural effusion, or pericardial effusion with symptoms and requiring intervention;
9. Esophageal or gastric varices requiring immediate intervention;
10. Not eligible to participate in this study at the discretion of the investigator;
11. Do not have adequate treatment washout period before study drug administration. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 24 months
  Occurrence and severity of adverse events (AEs), with severity determined by NCI CTCAE v5.0 criteria
Number of subjects with clinically significant changes in physical examination results | 24 months
  Clinically significant abnormal physical examination findings reported by the investigator.
Number of subjects with clinically significant changes in vital signs | 24 months
  Vital signs including body temperature, pulse, respiratory rate, SpO2 and blood pressure
MTD or RP2D of IBI3001 Number of subjects with dose-limiting toxicities (DLTs) | 24 months
  Dose limiting toxicity (DLT) to establish MTD or RP2D

SECONDARY OUTCOMES:
Plasma concentration (Cmax) of IBI3001 | 24 months
  Plasma concentration of IBI3001 for single and multiple doses.
Area under the curve (AUC) of IBI3001 | 24 months
  AUC of IBI3001 for single and multiple doses
Time to maximum concentration (Tmax) of IBI3001 | 24 months
  Tmax of IBI3001 for single and multiple doses.
Clearance (CL) of IBI3001 | 24 months
  Clearance of IBI3001 from the plasma
Volume of distribution (V) of IBI3001 | 24 months
  Apparent volume of distribution of IBI3001
Half-life (T1/2) of IBI3001 | 24 months
  T1/2 of IBI3001 for single and multiple doses
Immunogenicity of IBI3001 | 24 months
  Incidence of anti-drug (IBI3001) antibody
Objective response rate (ORR) | 24 months
  ORR as evaluated per the RECIST v1.1 criteria
Duration of response (DoR) | 24 months
  DoR as evaluated per the RECIST v1.1 criteria
Disease control rate (DCR) | 24 months
  DCR as evaluated per the RECIST v1.1 criteria
Time to response (TTR) | 24 months
  TTR as evaluated per the RECIST v1.1 criteria
Progression free survival (PFS) | 24 months
  PFS as evaluated per the RECIST v1.1 criteria
Overall survival (OS) | 24 months
  Overall survival.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (2):
  - Wollongong Public, Wollongong, New South Wales
  - Cancer Research SA, Adelaide, South Australia
- China (3):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No